CLINICAL TRIAL: NCT04403997
Title: Virtual Chromoendoscopy With Second Generation NBI (HQ190) vs Chromoendoscopy in Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, María Dolores Martín Arranz, PhD, Principal Investigator, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NBICromo
Record Dates: First submitted 2020-05-21; First posted 2020-05-27 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Chromoendoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chromoendoscopy with methylene blue 0.1% (Active Comparator): Once the cecum is reached, a spray catheter is introduced through the working channel and the dye, a 0.1% methylene blue solution, is applied.
  Interventions: Procedure: Chromoendoscopy
- Virtual Chromoendoscopy with NBI with HQ190 endoscopes (Experimental): Intubation is done with normal white light. Once the cecum is reached, the removal will be done in NBI mode
  Interventions: Procedure: Chromoendoscopy

INTERVENTIONS:
Procedure: Chromoendoscopy — Chromoendoscopy is an endoscopic technique used in the follow-up of inflammatory bowel disease of long evolution. Chromoendoscopy, through the application of specific dyes used directly on the intestinal mucosa, promotes the visualization of mucosal lesions.

SUMMARY:
Study to compare the detection of neoplastic lesions between chromoendoscopy and NBI

DETAILED DESCRIPTION:
Single-blind (patient) randomized study to compare detection of neoplastic lesions between chromoendoscopy and NBI.

Patients with Inflammatory Bowel Disease who are to undergo chromoendoscopy according to usual clinical criteria will be included. The endoscopic procedure is similar to the one usually performed. All patients will undergo colonoscopy according to the usual procedure, with Olympus HQ190 series endoscopes, with the same bowel preparation. During intubation, the faecal remains will be thoroughly washed.

Patients will be randomly assigned to one of the two techniques: Chromoendoscopy with 0.1% methylene blue or New generation NBI with Near focus.

Biopsies will be taken of all those lesions detected, instead of random biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of Inflammatory Bowel Disease with indication to undergo chromoendoscopy

Exclusion Criteria:

* Patients who are not trained to understand the nature of the study, the procedures to be followed or are not able to sign an informed consent
* Known allergy or intolerance to methylene blue
* Pregnant or lactating women
* Personal history of colorectal cancer
* Ulcerative colitis active more than 20 cm from the anal verge
* Patients with known G6PD deficiency
* Severe kidney failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-02-25 (Estimated)

PRIMARY OUTCOMES:
Lesions detected | Baseline
  Total number of IBD dysplastic lesions detected by the use of NBI virtual chromoendoscopy versus conventional chromoendoscopy

SECONDARY OUTCOMES:
Detection rate of dysplastic lesions | Baseline
  Number of patients with at least one dysplastic lesion
Non-dysplastic lesions | Baseline
  Assess the number of non-dysplastic lesions detected with both methods
Ratio of neoplastic lesions/total lesions | Baseline
  Compare the ratio of neoplastic lesions/total lesions between both groups
Total endoscopy time | Baseline
  The total endoscopy time is counted from the introduction of the endoscope in the patient until its complete removal
Removal time | Baseline
  Withdrawal time is counted from the time the cecum is reached to the completion of the test, including time spent on staining, biopsy or polypectomy
Near Focus ability | Baseline
  Assess Near Focus ability to optically differentiate dysplastic from non-dysplastic lesions
Number of biopsies | Baseline
  Number of biopsies taken in the different groups

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Martín Arranz, PhD, Principal Investigator — Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No